CLINICAL TRIAL: NCT06884449
Title: A Randomized, Double-Blind, Parallel, 3-Arm, Placebo-Controlled Study Evaluating the Effects of Arrabina P on Satiety in Healthy Adults
Brief Title: A Placebo-Controlled Study Evaluating the Effects of Arrabina P on Satiety in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comet Bio Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C02-24-01-T0076
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Satiety; Appetite Regulation; Weight Control
Keywords: Satiety; Appetite; Weight Management

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Parallel, 3-Arm, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Not Active Powder per sachet
  Interventions: Other: Placebo
- Arrabina P Prebiotic 5.0 g (Experimental): Active Arrabina P Prebiotic 5.0 g fiber per sachet
  Interventions: Dietary Supplement: Arrabina P Prebiotic 5.0 g
- Arrabina P Prebiotic 3.5 g (Experimental): Active Arrabina P Prebiotic 3.5 g fiber per sachet
  Interventions: Dietary Supplement: Arrabina P Prebiotic 3.5 g

INTERVENTIONS:
Dietary Supplement: Arrabina P Prebiotic 5.0 g — Active Powder
  Arms: Arrabina P Prebiotic 5.0 g
Dietary Supplement: Arrabina P Prebiotic 3.5 g — Active Powder
  Arms: Arrabina P Prebiotic 3.5 g
Other: Placebo — Placebo Powder
  Arms: Placebo

SUMMARY:
This study is being conducted to assess the effects of a prebiotic product, Arrabina P, on appetite in healthy adults. The goal is to see if this product can help with appetite regulation, support gut health, and support weight management.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel, 3-arm, placebo-controlled study to assess the effects of Arrabina P Prebiotic on satiety in healthy adults. The primary goal of this study is to assess how two different doses of Arrabina P affect self-reported appetite. Secondary goals include evaluating weight control, eating behaviors, mood, sleep quality, and memory. The product is expected to support beneficial gut bacteria, help maintain lipid levels, and promote digestive comfort and appetite regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male and female participants who are between 18 - 65 years of age (inclusive).
2. Have a body mass index (BMI) range of 25.0 - 29.9 kg/m2 (inclusive).
3. Female participants must meet one of the following criteria:

   * Have a regular menstrual cycle, defined as a consistent cycle length of 24-32 days for participants in the main group and 26-32 days for participants in the subgroup and demonstrated during the screening period
   * No longer menstruate due to medication (e.g., those taking birth control shots like Depo-Provera®)
   * No longer menstruate due to being postmenopausal, surgical removal of ovaries, or medically documented ovarian failure
4. Have the habit of consuming food in the morning daily, and agree to fully consume a standardized high-carbohydrate breakfast within 15 minutes at Visit 2, Visit 3 and Visit 4.
5. Have veins suitable for repeated blood sampling in subgroup only.
6. Have maintained dietary habits and lifestyle within 3 months prior to screening and willing to maintain their habitual diets and lifestyle throughout the study.
7. Agree to follow the restrictions on concomitant treatments as listed
8. Willing and able to adhere to the requirements and restrictions of this study, willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study.
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
3. Have Type I diabetes or Type II diabetes, high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or uncontrolled thyroid disease ("uncontrolled" defined as being unmedicated, have an unstable use of medication within 3 months prior to screening, or have a stable use of medication for 3 months but still have uncontrolled conditions).
4. Current high fiber intake (estimated to be ≥ 30 g per day as estimated by a questionnaire at screening).
5. Currently participating in a weight management program or on a specific diet (e.g., Atkins, keto, intermittent fasting, etc.), or participated in a weight management program with its completion occurred within 3 months prior to baseline.
6. Experienced a change in body weight of ±4.5 kg (10 lbs.) over the 3 months prior to baseline.
7. Have eating disorder(s) (e.g., bulimia, binge eating disorder, etc.).
8. Have medical condition(s) known to manifest gastrointestinal symptoms (e.g., irritable bowel syndrome, endometriosis, etc.).
9. Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).
10. Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).
11. Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer) with recovery occurred within 5 years before the screening visit.
12. Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, bipolar disorder, schizophrenia, etc.).
13. Reports a clinically significant illness during the 28 days before the first dose of study product.
14. Major surgery in 3 months prior to screening or planned major surgery during the study.
15. Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program) or use that to the opinion of the investigator may be of a concern for the study.
16. Currently, or plan to, live in the same household with another participant in the current study during the study period.
17. Current enrolment or past participation in another study with any product(s) with at least one active ingredient within 28 days before first dose of study product or longer, if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
18. Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 4
  Change from baseline to Week 4 in incremental area under the curve (iAUC) of the following self-reported appetite sensations, with each sensation measured using a 100 mm visual analogue scale (VAS) over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Hunger.
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 4
  Change from baseline to Week 4 in incremental area under the curve (iAUC) of the following self-reported appetite sensations, with each sensation measured using a 100 mm visual analogue scale (VAS) over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Fullness
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 4
  Change from baseline to Week 4 in incremental area under the curve (iAUC) of the following self-reported appetite sensations, with each sensation measured using a 100 mm visual analogue scale (VAS) over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Satiation
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 4
  Change from baseline to Week 4 in incremental area under the curve (iAUC) of the following self-reported appetite sensations, with each sensation measured using a 100 mm visual analogue scale (VAS) over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Prospective food consumption

SECONDARY OUTCOMES:
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 12
  Change from baseline to Week 12 in iAUC of the following self-reported appetite sensations, with each sensation measured using a 100 mm VAS over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Hunger
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 12
  Change from baseline to Week 12 in iAUC of the following self-reported appetite sensations, with each sensation measured using a 100 mm VAS over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Fullness
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 12
  Change from baseline to Week 12 in iAUC of the following self-reported appetite sensations, with each sensation measured using a 100 mm VAS over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Satiation
To evaluate the effect of TP at two dose levels on appetite control, compared to placebo | Week 12
  Change from baseline to Week 12 in iAUC of the following self-reported appetite sensations, with each sensation measured using a 100 mm VAS over 4 hours after the consumption of a standardized high-carbohydrate breakfast - Prospective food consumption
To evaluate the effect of TP at two dose levels on body weight, compared to placebo | Week 12
  Percent change from baseline to Week 12 in body weight
To evaluate the effect of TP at two dose levels on eating behaviours, compared to placebo | Week 4
  Change from baseline to Week 4 in eating behaviors as assessed by the following questionnaires 2 hours after the consumption of a standardized high-carbohydrate breakfast - Three-Factor Eating Questionnaire (TFEQ)
To evaluate the effect of TP at two dose levels on eating behaviours, compared to placebo | Week 12
  Change from baseline to Week 12 in eating behaviors' as assessed by the following questionnaires 2 hours after the consumption of a standardized high-carbohydrate breakfast - Three-Factor Eating Questionnaire (TFEQ)
To evaluate the effect of TP at two dose levels on eating behaviours, compared to placebo | Week 4
  Change from baseline to Week 4 in eating behaviors' as assessed by the following questionnaires 2 hours after the consumption of a standardized high-carbohydrate breakfast - Food Craving Questionnaire-Trait (FCQ-T)
To evaluate the effect of TP at two dose levels on eating behaviors, compared to placebo | Week 12
  Change from baseline to Week 12 in eating behaviors' as assessed by the following questionnaires 2 hours after the consumption of a standardized high-carbohydrate breakfast - Food Craving Questionnaire-Trait (FCQ-T)
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 4
  Change from baseline to Week 4 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Total Cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 12
  Change from baseline to Week 12 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Total Cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 4
  Change from baseline to Week 4 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: High-density lipoprotein (HDL) cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 12
  Change from baseline to Week 12 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: High-density lipoprotein (HDL) cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 4
  Change from baseline to Week 4 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Low-density lipoprotein (LDL) cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 12
  Change from baseline to Week 12 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Low-density lipoprotein (LDL) cholesterol
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 4
  Change from baseline to Week 4 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Triglycerides
To evaluate the effect of TP at two dose levels on blood lipid biomarkers, compared to placebo | Week 12
  Change from baseline to Week 12 in the following blood lipid biomarkers in fasting blood samples with each dose level of TP or placebo: Triglycerides
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Bifidobacteriaceae (B.longum) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Bifidobacteriaceae (B.longum) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Bifidobacteriaceae (B. bifidum) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Bifidobacteriaceae (B. bifidum) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Prevotellaceae (P. copri) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Prevotellaceae (P. copri) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Bacteriodes (C. cellulosilyticus) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Bacteriodes (C. cellulosilyticus) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Bacteriodes (B.thetaiotaomicron) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Bacteriodes (B.thetaiotaomicron) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Bacteriodes (B. intestinalis) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Bacteriodes (B. intestinalis) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Lactobacillaceae (Lactobacillus) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Lactobacillaceae (Lactobacillus) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Ruminococceae (F. prausnitzzi) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Ruminococceae (F. prausnitzzi) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Lachnospiraceae (R. hominis) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Lachnospiraceae (R. hominis) as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 4
  Change from baseline to Week 4 stool sample in the abundance of the following beneficial microbes: Akkermansia spp as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on microbiota composition, compared to placebo | Week 12
  Change from baseline to Week 12 stool sample in the abundance of the following beneficial microbes: Akkermansia spp as assessed by 16s RNA sequencing
To evaluate the effect of TP at two dose levels on gastrointestinal health, compared to placebo | Week 4
  Changes from baseline to Week 4 in gastrointestinal symptoms rating scales (GSRS)
To evaluate the effect of TP at two dose levels on gastrointestinal health, compared to placebo | Week 12
  Changes from baseline to Week 12 in gastrointestinal symptoms rating scales (GSRS)
To evaluate the effect of TP at two dose levels on mood, compared to placebo | Week 4
  Changes from baseline to Week 4 in mood state as assessed by the Brunel Mood Scale Questionnaire (BRUMS-24) total mood disturbance score and sub-scales
To evaluate the effect of TP at two dose levels on mood, compared to placebo | Week 12
  Changes from baseline to Week 12 in mood state as assessed by the Brunel Mood Scale Questionnaire (BRUMS-24) total mood disturbance score and sub-scales
To evaluate the effect of TP at two dose levels on sleep quality, compared to placebo | Week 4
  Changes from baseline to Week 4 in sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI)
To evaluate the effect of TP at two dose levels on sleep quality, compared to placebo | Week 12
  Changes from baseline to Week 12 in sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI)
To evaluate the effect of TP at two dose levels on memory, compared to placebo | Week 4
  Changes from baseline to Week 4 in memory as assessed by Multifactorial Memory Questionnaire (MMQ)
To evaluate the effect of TP at two dose levels on memory, compared to placebo | Week 12
  Changes from baseline to Week 12 in memory as assessed by Multifactorial Memory Questionnaire (MMQ)
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial glucose and insulin response, compared to placebo | Week 4
  Changes from baseline to Week 4 in the postprandial profile of glucose and insulin over 4 hours after a standardized high-carbohydrate breakfast with each dose level of TP or placebo

OTHER OUTCOMES:
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 4
  Changes from baseline to Week 4 in serum lipopolysaccharide binding protein (LBP), with each dose level of TP or placebo
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 12
  Changes from baseline to Week 12 in serum lipopolysaccharide binding protein (LBP), with each dose level of TP or placebo
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 4
  Changes from baseline to Week 4 in serum zonulin, with each dose level of TP or placebo
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 12
  Changes from baseline to Week 12 in serum zonulin, with each dose level of TP or placebo
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 4
  Changes from baseline to Week 4 and in fecal calprotectin, with each dose level of TP or placebo
To evaluate the effect of TP at two dose levels on gut permeability, compared to placebo | Week 12
  Changes from baseline to Week 12 and in fecal calprotectin, with each dose level of TP or placebo
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Vitals: Heart rate in beats per minute (bpm)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Vitals: Blood Pressure in mmhg
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Anthropometrics - Weight in kilograms (Kg)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Anthropometrics: Body Mass Index (Weight in kilograms (Kg) divided by the square of height in meters (m2)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Hemoglobin (g/dl)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Hematocrit (%)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Red Blood Cells (RBC) in million cells/mcL
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Red Blood Cell Distribution Width (RDW) in fL
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Mean Corpuscular Volume (MCV)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Mean Corpuscular Hemoglobin (MCH)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Mean Corpuscular Hemoglobin Concentration(MCHC)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: White Blood Cells (WBC) and differential (abs)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Platelet count
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Mean Platelet Volume (MPV)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Blood urea nitrogen (BUN)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Creatinine
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Bilirubin total
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Alkaline phosphatase
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: AST
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: ALT
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Albumin
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Total protein
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Sodium
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Potassium
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Estimated glomerular filtration rate (eGFR)
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Globulin
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Laboratory blood tests. Fasting blood samples will be collected to assess for changes in: Chloride
To assess the safety and tolerability of the TP in healthy participants | Week 12
  Reports of adverse events will be collected and compared between the TP and placebo group
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Acetic Acid will be quantified using GC-MS analysis
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Propionic acid will be quantified using GC-MS analysis
Subgroup only:To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Butyric acid will be quantified using GC-MS analysis
Subgroup only:To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Valeric acid will be quantified using GC-MS analysis
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Isovaleric acid will be quantified using GC-MS analysis
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Caproic acid will be quantified using GC-MS analysis
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial short-chain fatty acid (SCFA) blood profiles | Week 4
  Change from baseline to Week 4 in postprandial profile of the following SCFA over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Heptanoic acid will be quantified using GC-MS analysis
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial appetite regulating hormone response, compared to placebo | Week 4
  Change from baseline and Week 4 in postprandial profile of the following hormones over the following specified hours after the consumption of a standardized high-carbohydrate breakfast:
  Over 4 hours: Total Glucagon-like peptide-1 (GLP-1)
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial appetite regulating hormone response, compared to placebo | Week 4
  Change from baseline and Week 4 in postprandial profile of the following hormones over the following specified hours after the consumption of a standardized high-carbohydrate breakfast:
  Over 4 hours: Peptide YY (PYY)
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial appetite regulating hormone response, compared to placebo | Week 4
  Change from baseline and Week 4 in postprandial profile of the following hormones over the following specified hours after the consumption of a standardized high-carbohydrate breakfast:
  Over 2 hours: Cholecystokinin (CCK)
Subgroup only: To evaluate the effect of TP at two dose levels on postprandial inflammatory response, compared to placebo in a subgroup of participants | Week 4
  Changes from baseline to Week 4 in serum IL-6 response over 4 hours after the consumption of a standardized high-carbohydrate breakfast
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: p-Hydroxyphenyllactic acid
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: caffeicacid, methylcaffeate
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast:
  (E)-Osmundacetone, homovanillic acid, 3,4-Dimethoxyphenylacetic
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast:
  acid/Dihydroferulic acid, 3-hydroxyphenylacetic acid
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Acetylagmatine
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: N-acetylputrescine, N-acetylcadaverine
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: Stachydrine
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: 2-hydroxyvaleric acid
Subgroup only: To evaluate the effect of TP at two dose levels on gut metabolomics in blood, compared to placebo in subgroup of participants | Week 4
  Change from baseline to Week 4 in the following gut microbial metabolites over 4 hours after the consumption of a standardized high-carbohydrate breakfast: 5-aminolevulinic acid 2-hydroxyisocaproic acid

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Richard, Study Director — Comet Biorefining Inc.
Locations (3):
- United States (3):
  - Indago Research Health Center,Inc., Hialeah, Florida
  - Vantage Clinical Trials, LLC, Tampa, Florida
  - Boston Clinical Trials - Alcanza, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No